CLINICAL TRIAL: NCT03734354
Title: A Single-center, Open-label Study Evaluating the Pharmacokinetics, Tolerability and Safety of Single Dose Oral Brexpiprazole Tablets in Healthy Chinese Subjects
Brief Title: The Pharmacokinetics, Tolerability and Safety of Brexpiprazole in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 331-403-00024
Record Dates: First submitted 2018-11-02; First posted 2018-11-07 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2020-07

CONDITIONS: Health
MeSH Terms: interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 mg dosing group (Experimental): Dosing group 1, single/oral/with fasting, Brexpiprazole 1.0 mg, 1 tablets
  Interventions: Drug: Brexpiprazole
- 2 mg dosing group (Experimental): Dosing group 2, single/oral/with fasting, Brexpiprazole 1.0 mg, 2 tablets
  Interventions: Drug: Brexpiprazole
- 4 mg dosing group (Experimental): Dosing group 3, single/oral/with fasting, Brexpiprazole 1.0 mg, 4 tablets
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Brexpiprazole , single/oral/with fasting
  Other Names: Brex

SUMMARY:
This study is a single-center, open-label study evaluating the pharmacokinetics, tolerability and safety of single dose oral brexpiprazole tablets in healthy Chinese subjects. A total of 30 healthy adult subjects are to be enrolled into the study. Three dose groups will be set up, with about 10 subjects in each dose group. Subjects will enter 1 mg, 2 mg and 4 mg dose groups in sequence.

DETAILED DESCRIPTION:
A total of 30 healthy adult subjects are to be enrolled into the study. Three dose groups will be set up, with about 10 subjects in each dose group. Subjects will enter 1 mg, 2 mg and 4 mg dose groups in sequence.

After the clinical trial responsible physicians obtain the informed consent forms from subjects, the subjects will be screened 14 days to 1 days prior to taking the study drug (D-14~D-1).

One day prior to dosing in each group (D-1), the included subjects are hospitalized On the next day (D1), after completed the hospitalization inspection, eligible subjects will be assigned subject numbers to start with the first dose, complete corresponding examination, stay in hospital for observation and be discharged on Day 4 of medication. On days 6, 8, 10, 12 blood samples are collected and safety evaluation will be performed. Telephone follow-up will be performed on day Day31.

Blood samples are collected to determine and evaluate blood concentrations of Brexpiprazole and its main metabolite DM-3411 before dosing, and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264 hours after dosing, with 18 sampling points in total.

ELIGIBILITY:
Inclusion Criteria:

* 1. Sign the informed consent form
* 2.At the age of 18~45 years old (including upper and lower limits) when signing the informed consent form.
* 3.Body weight of not less than 50kg, BMI 19 ~ 24kg/m2 (including the upper and lower limits) [ body mass index (BMI) = body weight (kg) / height2 (m2)].

Exclusion Criteria:

* 1. Participated in any interventional clinical trial within 12 weeks prior to enrollment.
* 2.Drug abuse in the past 2 years or a history of abuse
* 3.Drinking alcohol more than 2 unit per day (1 unit= 360 ml beer , or 45 ml 4.0% alcohol, or 150 ml liquor, or 50 ml wine ) 6 months before the screening, or subjects can not stop drinking during the hospitalization

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-07 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
The peak concentration (Cmax) after the first administration | 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264 hours
  The peak concentration (Cmax) of Brexipiprazole and the metabolite DM-3411 after administration
The peak time (Tmax) after the first administration | 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264 hours
  The peak-time of Brexipiprazole and the metabolite DM-3411 on the first day after administration are calculated.
Area under the plasma concentration-time curve (AUC0-264h) | 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264 hours
  The area under the plasma concentration-time curve of Brexipiprazole after administration are calculated.
Half time after the first administration | 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264 hours
  The half time of Brexipiprazole after administration are calculated.
Apparent clearance after the first administration | 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264 hours
  To assess the apparent clearance after administration (CL/F) of Brexipiprazole after the first administration
Proportional dose-response relationship between pharmacokinetic parameters Cmax and AUC of OPC-34712 | 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264 hours
  To assess the Proportional dose-response relationship between pharmacokinetic parameters Cmax and AUC of OPC-34712

SECONDARY OUTCOMES:
Blood pressure | 0, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264 hours
  To seeess blood pressure after administration of brexpiprazole
Heart rate | 0, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264 hours
  To seeess heart rate after administration of brexpiprazole
Body weight | 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264 hours
  To seeess Body weight after administration of brexpiprazole
12-lead ECG | 3, 6, 24, 72, 96, 120, 264 hours
  To seeess 12-lead ECG after administration of brexpiprazole
Blood biochemistry | 24, 96, 264 hours
  To seeess blood biochemistry after administration of brexpiprazole
Blood routine | 24, 96, 264 hours
  To seeess blood routine after administration of brexpiprazole
urinary routine | 24, 96, 264 hours
  To seeess urinary routine after administration of brexpiprazole

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jiang, Master, Principal Investigator — Beijing Anding Hospital of Capital Medical University
Locations (1):
- Beijing Anding Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No